CLINICAL TRIAL: NCT06610825
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of Fam-Trastuzumab Deruxtecan-Nxki (T-DXd) as a Subsequent Line of Therapy in HER2-Positive Metastatic Castration-Resistant Prostate Adenocarcinoma
Brief Title: Castrate Resistant Prostate Cancer Enhertu Therapy
Acronym: CaRPET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Daiichi Sankyo (Industry); Cancer Research And Biostatistics (Unknown); Institute for Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1803020
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer Metastatic; Prostate Cancer; CRPC
Keywords: prostate cancer; metastatic prostate cancer; Enhertu; HER2 positive; Trastuzumab deruxtecan; crpc; phase 2
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enhertu for HER2 positive metastatic castrate resistant prostate cancer (Experimental)
  Interventions: Drug: Enhertu

INTERVENTIONS:
Drug: Enhertu — This is an open label, multi-center, single arm, phase II study designed to investigate the anti-tumor activity, efficacy and safety of Enhertu in HER2-positive metastatic castrate-resistant prostate cancer patients who progressed on androgen deprivation therapy and novel hormonal agents (such as Abiraterone and Enzalutamide), who also progressed, refused, or were not candidates to receive taxane-based chemotherapy.

SUMMARY:
Use of Enhertu as a Subsequent Line of Therapy in HER2-Positive Metastatic Castration-Resistant Prostate Adenocarcinoma.

DETAILED DESCRIPTION:
This Phase II clinical trial aims to evaluate the efficacy and safety of Enhertu in HER-2 positive mCRPC who have progressed on prior androgen deprivation therapy and novel hormonal agents, who are either not candidates for or have refused taxane based chemotherapy. Led by Dr. Maneesh Jain at the Washington DC VA, the open label multi center study will include 60 participants treated with Enhertu. Primary endpoints focus on objective response rates, while secondary measures include safety, progression-free survival, overall survival, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the prostate
* Diagnosis of mCRPC
* Documented progression on androgen deprivation and novel hormonal agents, with or without progression on taxane containing regimen
* Ongoing ADT to maintain serum testosterone levels below 50 ng/dL
* Formalin fixed paraffin embedded tumor tissue for HER2 immunohistochemistry
* Life expectancy 6 months
* ECOG 0 or 1
* LVEF at least 50%
* Adequate Blood Clotting function
* Adequate Organ and Bone Marrow function
* Adequate Renal function
* Adequate Hepatic function

Exclusion Criteria:

* History of interstitial lung disease or pneumonitis requiring steroids
* Significant coronary vascular disease
* Previous exposure to HER2 targeted therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  Objective Response Rate by local review, combining radiographic and biochemical responses

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
Overall Survival | 2 years
Disease Control Rate | 2 years
Duration of Response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maneesh Jain, MD, Study Chair — Washington DC VA Medical Center; Eric Knoche, MD, Principal Investigator — VA St. Louis Healthcare System; Suman Kambhampati, MD, Principal Investigator — VA Kansas City; Julie Graff, MD, Principal Investigator — Portland VA Medical Center; Bruce Montgomery, MD, Principal Investigator — VA Puget Sound HCS; David Kosoff, MD, Principal Investigator — Wisconsin VA Medical Center; Karan Jatwani, MD, Principal Investigator — George Washington University Cancer Center; Kerry Schaffer, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Washington DC VAMC, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajendran R, Lap CJ, Madapoosi S, Heiraty A, Estephan F, Hahn W, Poudel A, Nava VE, Subrahmanyam R, Jain M. Clinical response to novel combination of trastuzumab deruxtecan and abiraterone in HER2-expressing metastatic castration-resistant prostate cancer. Oncologist. 2025 Sep 1;30(9):oyaf207. doi: 10.1093/oncolo/oyaf207. PMID 40638235
- [Background] Lap CJ, Rajendran R, Martin JM, Uppal M, Escobar A, Heiraty AM, Estephan F, Hahn W, Subrahmanyam R, Nava VE, Jain M. Response of Human Epidermal Growth Factor Receptor 2-Expressing Prostate Cancer to Trastuzumab Deruxtecan. Ann Intern Med. 2024 Dec;177(12):1738-1741. doi: 10.7326/ANNALS-24-01409. Epub 2024 Nov 5. No abstract available. PMID 39496182
- [Background] Estephan F, Lap CJ, Banagan J, Antonio M, Liu S, Diao G, Rozalen AZ, Rajendran R, Krasnow S, Subrahmanyam R, Nava VE, Jain M. The prevalence and clinical significance of HER2 expression in prostate adenocarcinoma. Ann Diagn Pathol. 2023 Dec;67:152219. doi: 10.1016/j.anndiagpath.2023.152219. Epub 2023 Oct 20. PMID 38622987
- See also: Enhertu Drug Information — https://www.enhertu.com/